CLINICAL TRIAL: NCT00249522
Title: Vouchers vs. Prizes for Methadone Patients
Brief Title: Vouchers vs. Prizes for Methadone Patients - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: UConn Health (Other)
Responsible Party: Nancy Petry, Ph.D., UConn Health Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-13444-1; R01-13444-1
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-05

CONDITIONS: Substance Abuse
Keywords: contingency management; substance abuse treatment
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Contingency management

SUMMARY:
The purpose of this study is to compare voucher-based contingency management (CM) procedures to a lower-cost CM system that provides opportunities to win prizes. Cocaine-dependent outpatients are randomly assigned to (a) standard treatment, (b) standard treatment plus voucher CM for abstinence, defined by negative breath and urinalysis test results, or (c) standard treatment plus prize CM for abstinence, defined by negative breath and urinalysis test results. Urine and breath samples are collected 3x/week during Weeks 1-3, 2x/week during Weeks 4-6 and 1x/week during Weeks 7-12. Follow-up interviews are conducted 1,3,6 and 9 months following intake during which substance use and psychosocial functioning are assessed.

ELIGIBILITY:
Inclusion criteria:

* age > 18 years
* current DSM-IV diagnosis of cocaine dependence
* maintained on a stable dose of methadone for >1 month
* willing to sign informed consent
* English speaking

Exclusion criteria:

* serious, uncontrolled psychiatric illness (e.g., acute schizophrenia, bipolar disorder, or substantial suicide risk) on the basis of history or medical examination
* dementia (<23 on the Mini Mental State Exam)
* in recovery from pathological gambling as determined by DSM-IV criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2003-08; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Drug use | baseline and each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Petry, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States